CLINICAL TRIAL: NCT03731507
Title: KinectROM Application for Assessing Range of Motion in Upper and Lower Extremity: A Development and Validation Study
Acronym: KinectROM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saime Nilay Arman (Other)
Responsible Party: Sponsor-Investigator, Saime Nilay Arman, Assist.Prof., Istanbul University
Organization: Istanbul University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IstanbulUC
Record Dates: First submitted 2018-11-03; First posted 2018-11-06 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Range of Motion
Keywords: range of motion; upper extremity; lower extremity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Range of motion in upper extremity (Experimental): Assessment of shoulder: flexion/extension, abduction/adduction, internal/external rotation, elbow flexion/extension, hip: flexion/extension, abduction/adduction, internal/external rotation, knee: flexion/extension, ankle: dorsal flexion/plantar flexion
  Interventions: Device: Assessment of Range of Motion with Kinect Controller

INTERVENTIONS:
Device: Assessment of Range of Motion with Kinect Controller — A ROM measurement method called as KinectROM by us has been developed with Kinect Controller

SUMMARY:
The aim of the study is to investigate the validity and reliability of KinectROM application for objectively evaluating range of motion (ROM)

DETAILED DESCRIPTION:
The application KinectROM called has been developed for assessing ROM with Kinect controller by our team. So, shoulder, elbow, knee, hip and ankle ROM measurements will be made with universal goniometer and developed KinectROM application.

ELIGIBILITY:
inclusion Criteria: -Healthy individuals with 18-40 years

Exclusion Criteria:

-Have any limited extremity between the ages of 18-40 years.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Range of Motion | baseline
  ROM of shoulder, elbow, knee, hip and ankle will be made with universal goniometer and developed Kinect controller based measurement method.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)